CLINICAL TRIAL: NCT00201903
Title: The Roles of Tissue Factor in Malignant Gliomas
Status: Completed | Type: Observational
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Ontario Cancer Research Network (Network)
Other Study IDs: OCOG-2003-TFsubstudy
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2007-05

CONDITIONS: Venous Thromboembolism; Brain Tumors
Keywords: venous thromboembolism; brain tumours; glioma; tissue factor; blood coagulation; tumour progression; low molecular weight heparin
MeSH Terms: conditions — Venous Thromboembolism; Brain Neoplasms; Glioma; Thrombosis; Disease Progression

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To explore the relationship between tissue factor levels, tumour progression, activation of blood coagulation and venous thromboembolism with malignant glioma

DETAILED DESCRIPTION:
To explore the relationship between tissue factor levels, tumour progression, activation of blood coagulation and venous thromboembolism with malignant glioma

ELIGIBILITY:
Inclusion Criteria:

* participation in PRODIGE
* adult patients
* newly diagnosed, biopsy-confirmed grade III/IV malignant gliomas
* undergone craniotomy or stereotactic biopsy > 2 days and < 4 weeks before

Exclusion Criteria:

* have known hereditary thrombophilia
* are receiving experimental antiangiogenic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-01; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Lee, MD, Study Chair — Hamilton Health Sciences and McMaster University; William Geerts, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Mark Levine, MD, Principal Investigator — Ontario Clinical Oncology Group (OCOG); James Perry, MD, Principal Investigator — Toronto Sunnybrook Regional Cancer Centre; Janusz Rak, Principal Investigator — Hamilton Health Sciences and McMaster University; Jeffrey Weitz, MD, Principal Investigator — Hamilton Health Sciences and McMaster University
Locations (6):
- United States (2):
  - Henry Ford Hospital, Detroit, Michigan
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Toronto-Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario